CLINICAL TRIAL: NCT04095234
Title: Integrative Medicine for Pain in Patients With Advanced Cancer Trial (IMPACT)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-341
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Cancer Pain
Keywords: acupuncture; massage; IMPACT; 19-341
MeSH Terms: conditions — Cancer Pain; Tooth, Impacted | interventions — Acupuncture Therapy; Massage

STUDY DESIGN:
Intervention Model Description: Two-arm parallel (Acupuncture vs. Massage) randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Participants will receive up to 10 treatments in the first 10 weeks (+/- 4 days) and then receive monthly booster treatments (+/- 7 days) for up to 26 weeks.
  Interventions: Procedure: Acupuncture
- Massage (Active Comparator): Participants will receive up to 10 treatments in the first 10 weeks (+/- 4 days) and then receive monthly booster treatments (+/- 7 days) for up to 26 weeks.
  Interventions: Procedure: Massage

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture, a therapy of traditional Chinese medicine (TCM), involves penetrating the skin with thin, solid, metallic needles that are manipulated by hand or electrical stimulation. If the patient has an electronically charged device, they will not receive TENS stimulation.
  Arms: Acupuncture
Procedure: Massage — Massage, which involves the manual manipulation of muscles and other soft tissue areas of the body, is one of the earliest known forms of pain relief.
  Arms: Massage

SUMMARY:
The purpose of this study is to compare the long-term effectiveness of acupuncture versus massage in people living with advanced cancer. The study will test how the two approaches compare in helping people with pain and its related symptoms and improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or older
* Having a diagnosis of the following: stage III or IV lung cancer; any stage pancreatic cancer; unresectable cholangiocarcinoma; unresectable liver cancer; unresectable ampullary or peri-ampullary cancer or other stage IV gastrointestinal cancer; stage III or IV ovarian or fallopian tube cancers or other stage IV gynecologic cancer; stage IV breast cancer; stage III testicular cancer; stage IV genitourinary cancer; stage III or IV sarcoma; stage IV melanoma; stage III or IV head/neck cancer; stage IV endocrine cancer; or hematological malignancies (lymphoma, myeloma, and leukemia)
* Be ambulatory (Karnofsky functional score of ≥ 60)
* Having musculoskeletal pain, defined as regional (joints, extremities, back, neck) or more generalized (fibromyalgia or chronic widespread pain); Patients with a neuropathic component to their pain that involves the extremities or back will be eligible.
* Having musculoskeletal pain for at least 1 month
* Having had pain for at least 15 days in the preceding 30 days
* Having a pain rating of 4 or greater in worst pain on a 0-10 numerical rating scale in the preceding week
* Having an expected prognosis of greater than six months as judged by the treating oncologist or study physician

Exclusion Criteria:

* Having a platelet count <15,000
* Cognitive impairment precluding response to study assessments
* Unwilling to accept random assignment
* Unwilling to commit to the 26-week study time period
* Have non-musculoskeletal pain syndromes (headache, facial pain, chest pain, visceral abdominal pain) if these are the sole source of pain but can be present as co-morbid conditions as long as a patient has a primary musculoskeletal pain condition defined as above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Worst Pain | 26 weeks from randomization
  Worst Pain Item from the short-form Brief Pain Inventory (BPI). The short-form BPI will be used to quantify pain severity and pain interference. The BPI contains 4 pain severity items and 7 pain interference items, all rated on a scale from 0 to 10 (higher ratings indicate worse pain intensity/interference).

CONTACTS AND LOCATIONS:
Overall Officials: Jun J Mao, MD, MSCE, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Baptist Alliance MCI, Miami, Florida
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Booher A, Mao JJ, Muniz RC, Romero SAD, Li SQ, Lopez AM, Liou KT. Association between Hispanic Ethnicity and Greater Expectation of Benefit from Acupuncture or Massage for Pain in Cancer. J Immigr Minor Health. 2024 Oct;26(5):953-957. doi: 10.1007/s10903-024-01611-8. Epub 2024 Jul 8. PMID 38977653
- [Derived] Epstein AS, Liou KT, Romero SAD, Baser RE, Wong G, Xiao H, Mo Z, Walker D, MacLeod J, Li Q, Barton-Burke M, Deng GE, Panageas KS, Farrar JT, Mao JJ. Acupuncture vs Massage for Pain in Patients Living With Advanced Cancer: The IMPACT Randomized Clinical Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2342482. doi: 10.1001/jamanetworkopen.2023.42482. PMID 37962891
- [Derived] Romero SAD, Emard N, Baser RE, Panageas K, MacLeod J, Walker D, Barton-Burke M, Liou K, Deng G, Farrar J, Xiao H, Mao JJ, Epstein A. Acupuncture versus massage for pain in patients living with advanced cancer: a protocol for the IMPACT randomised clinical trial. BMJ Open. 2022 Sep 1;12(9):e058281. doi: 10.1136/bmjopen-2021-058281. PMID 36581960
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm